CLINICAL TRIAL: NCT00209170
Title: Depression-Diabetes Mechanisms: Urban African Americans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dominique Musselman, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00001092; R01MH069254-03 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Results first posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes; Depression
MeSH Terms: conditions — Diabetes Mellitus; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beating the Blues CBT + Escitalopram (Experimental): Subjects with type 2 diabetes will be randomized to Beating the Blues (computerized cognitive behavioral therapy) with the selective serotonin reuptake inhibitor (SSRI) antidepressant, escitalopram (10 mg taken orally once or twice daily) for 6 months
  Interventions: Behavioral: Beating the Blues; Drug: Escitalopram
- Beating the Blues CBT + Placebo (Active Comparator): Subjects with type 2 diabetes will be randomized to Beating the Blues (computerized cognitive behavioral therapy) with placebo (taken orally one to two tablets daily) for 6 months
  Interventions: Behavioral: Beating the Blues; Drug: Placebo

INTERVENTIONS:
Behavioral: Beating the Blues — Beating the Blues is a computerized cognitive behavioral therapy.
Drug: Escitalopram — Escitalopram is a selective serotonin reuptake inhibitor (SSRI) antidepressant. It's a 10 mg pill taken once or twice daily for 6 months.
  Other Names: Lexapro
  Arms: Beating the Blues CBT + Escitalopram
Drug: Placebo — A sugar pill taken as one to two tablets daily for 6 months.
  Arms: Beating the Blues CBT + Placebo

SUMMARY:
African-Americans suffer from increased prevalence of both type 2 diabetes and diabetes complications, reflecting a combination of psychobehavioral factors as well as metabolic dysfunction. In this process, depression may contribute to both the genesis of type 2 diabetes (through impact on neurohormonal activation, inflammatory mediators, and insulin resistance), and difficulties in management (through decreased adherence to diet plans, medication, and scheduled appointments). The preliminary data from the Grady Diabetes Clinic indicates that depression may be common in African-Americans with diabetes, that depression is a factor in non-adherence, and that non-adherence leads to poor glycemic control - a direct cause of diabetes complications. What is not known is: how treatment of depression could lead to both neurohormonal and psychobiological improvement, with improved patient adherence and glycemic control.

DETAILED DESCRIPTION:
To determine the psychobehavioral and neurohormonal mechanisms of effective treatment, the investigator will conduct a randomized, double-blind, placebo-controlled trial in patients with major depression, who will receive either: (i) computer-based cognitive behavioral therapy (CBT) program entitled "Beating the Blues" + placebo, or (ii) computer-based cognitive behavioral therapy (CBT) program entitled "Beating the Blues" + the SSRI antidepressant escitalopram. The investigator will assess (a) glycemic control (levels of glycated hemoglobin (HbA1c)), in relation to (b) adherence (keeping scheduled return appointments, diet, exercise, and glucose monitoring), (c) depressive symptoms (neurocognitive and neurobehavioral symptoms determined by self- and observer-rated scales), and (d) the four pathways of neurometabolic function.

Study visits will occur once a month for 6 months. Should patients report severe environmental stressors (such as marital conflict, loss of family member or job, being exposed to trauma), patients will be offered an intensification of their contact with study personnel, e.g. weekly contact by phone or "in-person" visits to see study personnel at the Grady Diabetes Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be English-speaking
* African American
* Have type 2 diabetes per American Diabetes Association criteria
* Patient's receiving care at Grady Hospital

Exclusion Criteria:

* Severely depressed (Hamilton Depression Rating Scale (HAM-D) ≥ 34
* Non - English speaking
* Women who are pregnant, women who will be breastfeeding during the study, and women of childbearing potential who are not practicing a reliable method of birth control.
* currently meet Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) criteria for:

  1. Bipolar Disorder
  2. Schizophrenia or any Psychotic Disorder
  3. Obsessive Compulsive Disorder
  4. Mental Retardation or any Pervasive Developmental Disorder or Cognitive Disorder.
  5. Personality Disorder of sufficient severity to interfere with their participation in the study
  6. Psychotic features or with history of Psychotic Disorder, as defined by DSM-IV
* Suicide risk, or have made serious suicide attempt in the past year
* Substance Abuse or Dependence (other than nicotine) during the six months preceding the first dose of double blind study medication
* Any malignancy (other than excised basal cell carcinoma), or any clinically significant hematological, endocrine, cardiovascular (including any rhythm disorder), renal, hepatic, gastrointestinal, or neurological disease. History of syndrome of inappropriate anti-diuretic hormone secretion.
* Diabetes due to: glucagonoma, pheochromocytoma or other endocrine neoplasm, drug induced diabetes, gestational diabetes, or those with established genetic defects of beta cell function.
* Medical conditions that will interfere with the HbA1c assay or if hospitalization is likely within two months (sickle cell anemia, hypersplenism)
* A history of diabetic ketoacidosis episode during the 6 months preceding the first dose of double-blind study medication.
* Uncontrolled diabetes as judged by the investigator defined as blood glucose greater than 400 on last two visits or patients whom suffered from diabetic ketoacidosis in the last month or have had 2 episodes in the last year.
* Autonomic or peripheral neuropathy that requires treatment
* At the first follow-up visit - Patients with systolic blood pressure greater than 180 mm Hg or less than 90 mm Hg or diastolic blood pressure greater than 105 mm Hg or less than 50 mm Hg
* Treatment with a depot neuroleptic during the last 6 months
* Patients who have been treated with any neuroleptic, antidepressant, or anxiolytic medication
* Participation in an investigational drug study within 1 month prior to study entry or who have received treatment with an investigational drug within 1 month or five half-lives, whichever is longer.
* Previous investigational study of escitalopram or previously treated with escitalopram in a dose and duration sufficient for therapeutic trial.
* History of hypersensitivity reaction to escitalopram or citalopram.
* Electroconvulsive therapy during the past 3 months
* Initiation or termination of behavior therapy or psychotherapy in the 3 months.
* Positive urine screening for alcohol, illicit drugs, or any prohibited medication

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique L Musselman, MD, MS, Principal Investigator — Emory University
Locations (1):
- Grady Hospital Diabetes Clinic, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consented 20 subjects, but 6 subjects were not randomized into treatment groups because they were lost to follow-up.
Groups:
- Beating the Blues CBT + Escitalopram: Subjects with type 2 diabetes randomized to Beating the Blues (computerized cognitive behavioral therapy) with the selective serotonin reuptake inhibitor (SSRI) antidepressant, escitalopram (10 mg taken orally once or twice daily) for 6 months
- Beating the Blues CBT + Placebo: Subjects with type 2 diabetes randomized to Beating the Blues (computerized cognitive behavioral therapy) with placebo (taken orally one to two tablets daily) for 6 months
Period: Overall Study
Arm/Group | Beating the Blues CBT + Escitalopram | Beating the Blues CBT + Placebo
Started | 7 | 7
Completed | 5 | 4
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beating the Blues CBT + Escitalopram | Beating the Blues CBT + Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Response of Participants, Defined by Change in the 21-item Hamilton Depression Rating Scale (HDRS) From Baseline to Week 24
Description: The 21-item HDRS measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 60, where higher scores indicate greater severity. The HDRS at week 24 was compared to the baseline HDRS and each participant's response was calculated using the below table:
  No Response = < 25% change in Depression Rating Scale Score Partial Responder =< 50% to >25% change in Depression Rating Scale Score Responder = 50% or greater change in Depression Rating Scale Score
Time Frame: Baseline, week 24
Population: Last Observation Carried Forward
Measure: Number; unit: participants
Arm/Group | Beating the Blues CBT + Escitalopram | Beating the Blues CBT + Placebo
Number analyzed (Participants) | 7 | 7
participants
  Response | 2 | 1
  Partial Response | 2 | 1
  No Response | 3 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data collected up to 6 months
Arm/Group | Beating the Blues CBT + Escitalopram | Beating the Blues CBT + Placebo
Serious Adverse Events (participants affected / at risk) | 1/7 | 2/7
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beating the Blues CBT + Escitalopram (N=7) | Beating the Blues CBT + Placebo (N=7)
Suicide attempt using insulin (Psychiatric disorders) | 0 (0) | 1 (1)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Beating the Blues CBT + Escitalopram (N=7) | Beating the Blues CBT + Placebo (N=7)
Chest tightness (Cardiac disorders) | 2 | 1
Orthostatic tachycardia (Cardiac disorders) | 1 | 2
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Sedation (Nervous system disorders) | 2 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 0
Sweating (Skin and subcutaneous tissue disorders) | 1 | 2
Weight gain (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Edema (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Frequent urination (Renal and urinary disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 5
Elevated blood pressure (Cardiac disorders) | 2 | 2
Insomnia (General disorders) | 3 | 1
Memory Difficulties (Nervous system disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Nose bleed (Ear and labyrinth disorders) | 0 | 1
Orthostatic hypotension (Cardiac disorders) | 1 | 2
Numbness (Musculoskeletal and connective tissue disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Sinus Congestion (Ear and labyrinth disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Tooth abscess (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyspnea (Cardiac disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No